CLINICAL TRIAL: NCT05492695
Title: TOGETHER STUDY: Tandem OnabotulinumtoxinA Galcanezumab Emerging Therapeutic Headache Elimination Research Study
Brief Title: Tandem OnabotulinumtoxinA Galcanezumab Emerging Therapeutic Headache Elimination Research Study
Acronym: TOGETHER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped from financial sponsor due to inability to enroll participants.
Sponsor: Diamond Headache Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5Q-US-X003
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Galcanezumab + BMPT (Active Comparator): * 240 mg of galcanezumab will be administered once as a loading dose at Visit 2, followed by monthly doses of 120 mg at Visits 3 and 4.
  * All participants will be required to continue BMPT. For consistency purposes visit 2/ randomization should be scheduled within +/- 3 days of subjects next Botox administration as part of BMPT.
  Interventions: Drug: Galcanezumab
- Placebo + BMPT (Placebo Comparator): • Galcanezumab matching placebo will be administered at Visits 2, 3 and 4.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Galcanezumab is a calcitonin-gene related peptide antagonist indicated in adults for the preventive treatment of migraine and the treatment of episodic cluster headache.
  Arms: Galcanezumab + BMPT
Other: Placebo — Galcanezumab' placebo. This is the same vehicle as the study intervention formulation but does not contain active galcanezumab-gnlm.
  Arms: Placebo + BMPT

SUMMARY:
This is a multicenter, double-blind, placebo-controlled study assessing the effectiveness of Galcanezumab as an add-on therapy for Migraine participants on a stable migraine prophylaxis regimen including Botox with or without one other migraine prophylaxis agent (BMPT), who have persistent unmet need. The study population will consist of approximately 150 participants ages 18-65 who report at least a 30% reduction in monthly migraine days from BMPT and still experience an average of ≥ 6 migraine days per month, following International Classification of Headache Disorders (ICHD-3) criteria. Subjects should be stable on at least 2, but no more than 8, consecutive injection cycles of Botox. Overall migraine day reduction will be assessed in the participants based on participant self-report (via daily electronic diaries) and medical record review.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate and sign informed consent;
2. Ability to understand informed consent and study procedures, including ability to use the electronic Daily Headache Diary;
3. In good general health based on investigator's judgment;
4. Must be between 18 to 65 years of age, inclusive, at time of Visit 1;
5. Reports having an average of > 6 migraine days per month, after at least 2 and up to 8 consecutive treatments of onabotulinumtoxinA at the time of screening, meeting the diagnostic criteria listed in the International Classification of Headache Disorders (ICHD-3);
6. Subject reports a > 30% decrease in the number of monthly migraine days from the onset of treatment with Botox (onabotulinumtoxinA);
7. Has a score on the Migraine Disability Assessment Questionnaire (MIDAS) >11 at screening;
8. During the baseline period reports >6 migraine days per month and < 25 days of head pain;
9. Onset of migraine before age 50;
10. Able to differentiate migraine from other primary headache types allowed in the study (e.g., tension-type headache);
11. Agrees to present for screening 28 days (± 3 days) prior to next anticipated Botox treatment, and to continue BMPT documented at screening for the rest of the study period. Subjects unwilling or unable to continue BMPT will not proceed through the study.;
12. Women may be included only if they have a negative pregnancy test at screening and baseline, are sterile, or postmenopausal. Women of childbearing potential (WOCBP) whose male partners are potentially fertile (i.e., no vasectomy) must use highly effective birth control methods for the duration of the study (i.e., starting at screening). Definitions of WOCBP, sterile and postmenopausal women, male contraception, and highly effective and acceptable birth control methods are to be determined based on investigator's judgment;
13. Demonstrated > 85% compliance the electronic Daily Headache Diary during 28-day run-in period (as defined as data entry on a minimum of 24 of the first 28 days of run-in period).

Exclusion Criteria:

1. Unable to understand the study requirements, the informed consent, or complete headache diaries as required per protocol;
2. Pregnant, actively trying to become pregnant, or breast-feeding;
3. Reports daily head pain during the month prior to screening;
4. Relevant history of substance abuse and/or dependence, in the opinion of the investigator;
5. History of impaired renal function that, in the investigator's opinion, contraindicates participation in this study;
6. Suffers from a serious illness, or an unstable medical condition, one that could require hospitalization, or could increase the risk of adverse events;
7. A psychiatric condition, in the opinion of the investigator, that may affect the interpretation of efficacy and safety data or contraindicates the participant's participation in the study;
8. Received nerve blocks or trigger point injections in the previous 8 weeks or plans to receive them during the study;
9. Exposure to biologics targeting the CGRP pathway in the previous 6 months or 5 half-lives, whichever is longer, or reports treatment with > 8 doses of small molecules targeting the CGRP pathway for acute abortive therapy in the last 30 days any CGRP blocker utilized for prevention of migraine is excluded from participation;
10. Has failed more than 3 classes of the following medications for the prevention of migraine due to a lack of efficacy (defined as no meaningful reduction in frequency of migraine days after an adequate trial of at least 2 months at generally accepted therapeutic doses), or >6 migraine preventative medications of any type, based on investigator's judgement

    1. Propranolol, metoprolol, atenolol, bisoprolol, timolol, or nadolol
    2. Topiramate
    3. Flunarizine
    4. Valproate or divalproex
    5. Amitriptyline or nortriptyline
    6. Venlafaxine or desvenlafaxine
    7. Lisinopril
    8. Candesartan
11. Received any investigational agents within 30 days prior to Visit 1;
12. Plans to participate in another clinical study at any time during this study;
13. History of medication overuse of opioids or butalbital (as defined by use ≥10 days per month) in previous 12 months or during run-in period; MOH (as defined by ICHD-3) with other medication types will be allowed but must be documented;
14. Use of more than 1 other medication, in addition to onabotulinumtoxinA for the prevention of migraine 12 weeks prior to screening or throughout the study;
15. Experienced a change in any concomitant migraine therapies in the12 weeks prior to screening or any non-migraine therapies which could confound assessment of response to IP in the opinion of the investigator;
16. Has a history of hyper-sensitivity reaction to any monoclonal antibody therapy or any component of galcanezumab injections;
17. Clinically relevant lab abnormalities at screening as determined by the investigator;
18. Clinically relevant or significant ECG abnormalities, including but not limited to ECG with QT interval corrected for heart rate (QTc) using Fridericia's correction formula (QTcF) > 500 msec; in the investigators opinion.
19. History of any of the following cardiovascular conditions:

    * Moderate to severe congestive heart failure (New York Heart Association class III or IV);
    * Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting;
    * Uncontrolled hypertension as defined by a confirmed systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
20. Active HIV or Hepatitis C infection;
21. Score of > 0 on question 9 of the Patient Health Questionnaire (PHQ-9) at any visit;
22. Have any other condition, in the judgment of the investigator, would make the participant unsuitable for inclusion, or would interfere with the participant participating in or completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Change in Monthly Migraine Days | Baseline to Treatment Month 3

SECONDARY OUTCOMES:
Change in Monthly Migraine days | Baseline to Treatment Months 1, 2, & 3
Change in Monthly Headache days | Baseline to Treatment Months 1, 2, & 3
Change in PROMIS Pain Interference scores | Baseline to Treatment Months 1, 2, & 3
Change in Functional Assessment of Migraine Scale - Research (FAMS-R) scores | Baseline to Treatment Months 1, 2, & 3
Change in Functional Assessment of Migraine Scale - Research Supplement (FAMS-RS) scores | Baseline to Treatment Months 1, 2, & 3
Change in Migraine Disability Assessment (MIDAS) scores | Baseline to Treatment Months 1, 2, & 3
Frequency of 50% Responders | Baseline to Treatment Months 1, 2, & 3
  50% Responders is defined as at least 50% reduction in number of monthly migraine days compared to baseline
Monthly Acute Migraine Medication use | Baseline to Treatment Months 1, 2, & 3

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Rhyne, MD, Study Director — Diamond Headache Clinic
Locations (1):
- Diamond Headache Clinic, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No